CLINICAL TRIAL: NCT06362044
Title: The Frequency of uMRD in Japanese Patients With CLL After 24 Months of Treatment With Venetoclax±Rituximab in the 2L+ in the Real-World Setting
Brief Title: A Study to Assess Frequency of Undetectable Minimal Residual Disease (uMRD) in Adult Participants With Chronic Lymphocytic Leukemia (CLL) Receiving Oral Venetoclax Tablets ± Intravenously (IV) Infused Rituximab in Routine Clinical Practice in Japan
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-120
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Venetoclax; Rituximab; ABT-199
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia (CLL) Participants: Participants will receive treatments for CLL in accordance with approved local label.

SUMMARY:
Most cases of Chronic lymphocytic leukemia (CLL) remain an incurable disease with the goal of therapy being to improve quality of life and to prolong survival. This study will evaluate the participant's related outcomes and experience of CLL in adult participants who are treated in the Japan.

Study participants will receive oral treatments of Venetoclax±Rituximab for CLL as prescribed by their study doctor in accordance with approved local label. Adult participants prescribed various treatments Venetoclax±Rituximab will be enrolled. Around 89 participants will be enrolled in the study in sites in Japan.

Participants will receive oral venetoclax tablets ± intravenously (IV) infused rituximab treatments for CLL according to the approved local label. The overall study duration will be 27 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with relapsed/refractory (2 Line [2L]+) chronic lymphocytic leukemia (CLL) in Japan based on International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria at the time of informed consent (IC).
* Treatment with Venetoclax±Rituximab for 24 months who are not treated with any other concurrent CLL treatment.
* Expected to visit the hospital at + 3 months after treatment with Venetoclax±Rituximab for 24 months.

Exclusion Criteria:

* No data on information on the start and end dates or continuation of treatment with Venetoclax.
* Participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with chronic lymphocytic leukemia (CLL) treated with Venetoclax±Rituximab and attend to a regular follow up visit at a Japanese participating hospital will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Undetectable Minimal Residual Disease (uMRD) | Up to 27 Months
  UMRD is defined as <10^-4 in peripheral blood (PB) assessed by flow cytometry (FCM).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- National Cancer Center Hospital East /ID# 265970, Kashiwa-shi, Chiba, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P24-120#additional-resources-section